CLINICAL TRIAL: NCT02626078
Title: Assessment of Food Practices by Residents in Nursing Homes, Study of Relationship Between Food Intake and Nutritional Status.
Brief Title: Assessment of Food Practices by Residents in Nursing Homes
Acronym: ARC2
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL14_0433
Record Dates: First submitted 2015-11-26; First posted 2015-12-10 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Malnutrition
Keywords: Malnutrition; Food practices; Elderly; Nursing Home; Aging; Nutritional status; Quality of life
MeSH Terms: conditions — Malnutrition | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observation and interview of residents: residents will be observed over lunch and an interview will be held with each resident after lunch
  Interventions: Other: observation and interview of residents

INTERVENTIONS:
Other: observation and interview of residents — Residents will be observed during lunch to evaluate their behavior, verbal interactions between residents. The food intake during 24 hours will be evaluated also. In an interview after lunch, the appreciation of the meal by residents will be assessed by a questionnaire and the score of the nutritional state will be defined.

SUMMARY:
Nutrition is an essential component of health and a key determinant of aging and quality of life of individuals. Malnutrition in the elderly is now recognized as a public health problem affecting nearly half of residents in nursing homes. The fight against malnutrition requires to rethink the meal in all its dimensions, beyond the nutritional needs. In order to improve practices of care at the elderly, the impact of environmental and social aspects of food in nursing homes has been assessed. The social environment and interactions during the meals are now identified as effective ways to stimulate food intake and increase feelings of well-being in the elderly.

The objectives of the study are to characterize the appreciation of food and social interactions during the meals and to study the relationships between the quality of food practices and nutritional status of the residents in nursing homes to improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Men or women living in nursing homes
* Person able to consent and understand the study
* Person able to converse in French, answer to a questionnaire
* Person feeding orally with or without assistance
* Person having lunch in community
* Availability of assessment criteria in the medical file

Exclusion Criteria:

* Person with cachexia syndrome
* Person with severe dementia (MMS <20)
* Dependent person (GIR score 1 and 2)
* Person with severe disorders of neurological origin swallowing
* Person under artificial nutrition (enteral, parenteral)
* Person with acute infectious disease
* Person with unstable medical or psychological conditions that could lead to be non receptive or uncooperative during the study or could compromise the security or the participation of the subject in the study
* Person under trusteeship or deprived of their liberty by judicial or administrative decision
* at the end of life

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The protocol will include 110 subjects recruited in nursing home in which they reside
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Assessment score of food practices | during lunch, an average of 30 minutes
  A questionnaire will be administered to the residents to target several criteria based on the assessment of the self-perception of the restaurant area, the hunger, the quality of food and services, the conviviality… A choice of four answers will be offered on each question to assess the level of appreciation of each criterion.

SECONDARY OUTCOMES:
Food intake (semi- quantitative estimation of the calorie and protein intakes). | 24 hours
  Visual estimation of the consumption of served portions, combined with the composition of each component of the 3 meals and snacks. The potential use of oral nutritional supplements will be included. Visual estimation of the consumption of portions shall be notified in a specific evaluation sheet (0, 25%, 50%, 75 % or 100% consumption of portions served) for each component of meal and snack.
Nutritional status | during the 30 minutes of the interview
  The mini nutritional assessment (MNA) will be completed for grading the nutritional state of the residents.
study the interactions developed during the meal between the subject and his entourage | during lunch, an average of 30 minutes
  A specific grid designed to easily capture different parameters characterizing the action of eating in community will be completed
health assessment of the resident at inclusion | at the inclusion visit
  a clinical examination will be made by the doctor

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Les Volubilis, Décines-Charpieu
  - Les Cristallines, Lyon
  - Les Amandines, Lyon
  - La Vérandine, Lyon
  - Castellane, Rillieux-la-Pape
  - Les Alizés, Saint-Priest
  - Les Althéas, Vaulx-en-Velin
  - Les Acanthes, Vaulx-en-Velin